CLINICAL TRIAL: NCT03938311
Title: Time Window for Early Mobilization in Improving Prognostic Outcomes in Patients With Acute Ischemic Stroke: an Investigator-Initiated Prospective Multicenter Randomized 3-Arm Clinical Trial
Brief Title: Time Window for Ischemic Stroke First Mobilization Effectiveness
Acronym: TIME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Stroke Databank Center (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Nanjing Tongren Hospital (Other); The First Affiliated Hospital of Soochow University (Other); Nanjing Jiangbei People's Hospital (Other); The First People's Hospital of Lianyungang (Other); The First Affiliated Hospital of Zhengzhou University (Other); Zibo Central Hospital (Other Government); Liaocheng People's Hospital (Other); Shandong Provincial Hospital (Other Government); Xingtai People's Hospital (Other); The First Hospital of Hebei Medical University (Other); Cangzhou Central Hospital (Other); Anhui Provincial Hospital (Other Government); The First Affiliated Hospital of Bengbu Medical University (Other); Jingmen No.1 People's Hospital (Other); Wuhan University (Other); Hainan General Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Shanghai Pudong Hospital (Other); Tianjin Medical University General Hospital (Other); Chongqing Three Gorges Central Hospital (Other); First Affiliated Hospital of Fujian Medical University (Other); First People's Hospital of Yulin (Other); First Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Xiao Lu,MD, Chief Physician, China Stroke Databank Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GN-2018R0010
Record Dates: First submitted 2019-04-27; First posted 2019-05-06 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Brain Ischemia; Stroke Rehabilitation
Keywords: Acute ischemic stroke; early rehabilitation; early mobilization; time window; multicenter randomized controlled trial
MeSH Terms: conditions — Brain Ischemia; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Patients with acute ischemic stroke fulfilling the inclusion and exclusion criteria will be randomly allocated to either either (1) the very early mobilization group in whichmobilization is initiated within 24 hours from stroke onset, (2) the early mobilization group in which mobilization begins between 24 and 72 hours poststroke, or (3) the late mobilization group in which mobilization is started after 72 hours poststroke.
Who Masked: Outcomes Assessor
Masking Description: Pre-admission trial assistants and medical staff aware of group allocation will not have contact with the patients. At each study site, a group of physiotherapists will be responsible for the interventions for all three study groups. Multi-disciplinary physicians, assessors, data analysts, and statisticians will be blinded to the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- very early rehabilitation (Experimental): early mobilization initiates within 24h from the onset of the disease
  Interventions: Other: early rehabilitation
- relative early rehabilitation (Experimental): early mobilization initiates between 24-72h from the onset of the disease
  Interventions: Other: early rehabilitation
- late mobilization group (Experimental): early mobilization initiates after 72h from the onset of the disease
  Interventions: Other: early rehabilitation

INTERVENTIONS:
Other: early rehabilitation — The three study groups share a same intervention protocol in addition to the initiation timing of intervention from the stroke onset. The frequency and intensity of the intervention is titrated according to functional activity baseline and monitored daily and adjusted with recovery. Encourage patients to move out of bed as soon as possible.
  Definition of bed movement: Encourage and help patients to perform functional actions, focusing on activities such as sitting, standing, walking out of the bed.

SUMMARY:
Early mobilization was thought to be effective in patients with acute ischemic stroke. As the essential component of stroke unit care, early mobilization has already been part of routine clinical practice. However, it is uncertain that which and when medical service focusing on functional recovery should be delivered after the emergency interventions for stroke. Besides, the optimal time window, for delivering early mobilization after acute ischemic stroke, has not been verified with strong evidence.

DETAILED DESCRIPTION:
The TIME Trial is a pragmatic, investigator-initiated, multi-center, randomized, 3-arm parallel group, clinical trial. This trial will be conducted in 57 general hospitals in mainland China affiliated with the China Stroke Databank Center and will enroll 6033 eligible patients with acute ischemic stroke. Participants will be randomly allocated to either (1) the very early mobilization group in whichmobilization is initiated within 24 hours from stroke onset, (2) the early mobilization group in which mobilization begins between 24 and 72 hours poststroke, or (3) the late mobilization group in which mobilization is started after 72 hours poststroke. The mobilization protocol is otherwise standardized and identical for each comparison group. Mobilization is titrated by baseline mobility level and progress of patients throughout the intervention period. The primary outcome is death or disability assessed with the modified Rankin scale at 3 months poststroke. Secondary outcomes include impairment score of the National Institutes of Health Stroke Scale, dependence in activities of daily living as measured using the modified Barthel Index, cognitive ability assessed with the Mini-Mental State Examination, incidence of adverse events, hospital length of stay, and total medical costs.

Study design: an Investigator-Initiated Prospective Multicenter Randomized 3-Arm Clinical Trial

Sample size: 1500 cases

ELIGIBILITY:
Inclusion Criteria:

* 1 diagnosed with ischemic stroke through anamnesis, clinical symptoms, and radiographic assessment;
* 2 aged 18 years or older;
* 3 of ischemic stroke within 12 hours before eligibility check;
* 4 able to verbally respond to the instructions;
* 5 with stable vital signs (systolic blood pressure 120-180 mmHg, heart rate 50-100/min, body temperature <37.5◦C, blood oxygen saturation >92%)
* 6MMSE score > 16;
* 7participation in the TIME Trial and sign the consent form.

Exclusion Criteria:

* 1 diagnosed with hemorrhagic stroke;
* 2 NIHSS score < 2;
* 3 pre-morbid modified Ranking Scale (mRS) score of 3-5;
* 4 refusing randomization;
* 5 having severe limb dysfunction or systemic diseases rendering them unable to cooperate in the mobilization intervention;
* 6 having severe cognitive and mental dysfunctions;
* 7 currently enrolled in another trial or having participated in a clinical trial within 6 months before stroke onset.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2019-08-13 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale | 3 months after the cerebrovascular accident/or the last time appeared normally
  modified Rankin Scale, to evaluate a subject's disability status. It's a rating data. The degrees range from 0 to 6, higher values represent a worse outcome and severe disability.

SECONDARY OUTCOMES:
Barthel Index | the total score of Barthel Index will be recorded 15days、1month、3 months、6months after the cerebrovascular accident/or the last time appeared normally
  ability of daily living, total scores range from 0 to 100, higher values represent a better outcome and independent living ability.
modified Rankin Scale | the total score of mRS will be recorded 15days、1month、6months after the cerebrovascular accident/or the last time appeared normally
  modified Rankin Scale, to evaluate a subject's disability status. It's a rating data. The degrees range from 0 to 6, higher values represent a worse outcome and severe disability.
MMSE | the total score of MMSE will be recorded 15days、1month、3 months、6months after the cerebrovascular accident/or the last time appeared normally
  Mini-mental State Examination. To evaluate a subject's mental state.The total score range from 0 to 30, higher values represent a better outcome.
NIHSS scores | the total score of NIHSS will be recorded15days、1month、6months after the cerebrovascular accident/or the last time appeared normally
  National Institute of Health stroke scale，total scores range from 0 to 42, higher values represent a better outcome.
Incidence of important medical events | The incidence of important medical events will be recorded 15days、1month、3 months after the cerebrovascular accident/or the last time appeared normally
  falls, trauma, fracture, syncope, epilepsy, pneumonia, atelectasis, venous thrombosis, pulmonary embolism, pressure sores, death, etc.
Hospital LOS | Hospital LOS will be recorded 3 months after the cerebrovascular accident/or the last time appeared normally
  length of stay in the acute hospital and in the rehabilitation hospital, and total hospital length of stay
Total medical cost | medical cost will be recorded 3 months after the cerebrovascular accident/or the last time appeared normally
  addition of the cost of each admission of the acute hospital and the rehabilitation hospital

OTHER OUTCOMES:
CBF | the count of CBF will be recorded 3months after the cerebrovascular accident/or the last time appeared normally
  cerebral blood flow
CBV | the count of CBV will be recorded 3months after the cerebrovascular accident/or the last time appeared normally
  cerebral blood volume
FA | 3months after the cerebrovascular accident/or the last time appeared normally
  fractional anisotropy, a outcome of diffusion tensor imaging
MD | 3months after the cerebrovascular accident/or the last time appeared normally
  mean diffusivity,a outcome of diffusion tensor imaging
rsFC | the rsFC description will be recorded by a radiologist 3months after the cerebrovascular accident/or the last time appeared normally
  resting-state functional connectivity

CONTACTS AND LOCATIONS:
Overall Officials: Lu Xiao, MD/PHD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University (Jiangsu Provincial People's Hospital), Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Zheng Y, Yan C, Shi H, Niu Q, Liu Q, Lu S, Zhang X, Cheng Y, Teng M, Wang L, Zhang X, Hu X, Li J, Lu X, Reinhardt JD; TIME Trial Collaboration Group. Time Window for Ischemic Stroke First Mobilization Effectiveness: Protocol for an Investigator-Initiated Prospective Multicenter Randomized 3-Arm Clinical Trial. Phys Ther. 2021 May 4;101(5):pzab038. doi: 10.1093/ptj/pzab038. PMID 33513232